CLINICAL TRIAL: NCT01021462
Title: An Open-Label, 2-Period, Pilot Study in Healthy Male Subjects to Evaluate the Use of a Graded Infusion of Intravenous Glucose in the Assessment of Insulin Secretion Rates
Brief Title: A Study to Evaluate the Use of a Graded Infusion of Intravenous Glucose in the Assessment of Insulin Secretion Rates (MK-0000-078)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0000-078; 078; 2009_695
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Period 1 + Period 2 (Experimental): graded infusion of intravenous glucose
  Interventions: Procedure: Comparator: graded infusion of intravenous glucose

INTERVENTIONS:
Procedure: Comparator: graded infusion of intravenous glucose — A stepwise graded infusion of glucose (20% dextrose [D20]) with a stable rate of infusion maintained for 40 minutes for each of 5 steps, with steps at 2,4,6,8 and 12mg/kg/min. Procedure will be identical in Period 1 and Period 2.

SUMMARY:
A two period pilot study to determine if a graded glucose infusion using a glucose (20% dextrose [D20]) intravenous infusion can be properly implemented and will be well tolerated in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is a non-smoker

Exclusion Criteria:

* Subject has a history of hypertension requiring treatment
* Subject has a history of cancer
* Subject's parents of siblings have a history of type 2 diabetes
* Subject is unable to refrain from the use of any prescription or non-prescription medication
* Subject consumes excessive amounts of alcohol or caffeine
* Subject has had major surgery, donated blood or participated in another investigational study in the past 4 weeks

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
proper implementation and tolerability of a grade glucose infusion using D20 intravenous infusion measured by glucose, insulin and C-peptide levels | 0-160 minutes after start of infusion

SECONDARY OUTCOMES:
beta-cell glucose sensitivity (slope of the relationship between insulin secretion rate and glucose) | 0-160 minutes after start of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC